CLINICAL TRIAL: NCT06789146
Title: Comparison of the Postoperative Analgesic Effects of Serratus Posterior Superior Intercostal Plane Block and Thoracic Paravertebral Block in Mastectomy Operations
Brief Title: Comparison of the Postoperative Analgesic Effects of SPSIPB and TPB in Mastectomy Operations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Atakan Sezgi, Principal İnvestigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AEŞH-EK-2025-07
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Mastectomy; Peripheral Nerve Block; Pain Management
Keywords: Mastectomy; Serratus Posterior Superior Intercostal Plane Block; Thoracic Paravertebral Block
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serratus posterior superior intercostal plane block (Active Comparator): After the patients are monitored and in the supine position, after appropriate field sterilization, a serratus posterior superior intercostal plane block will be performed on the patients using 30 ml of local anesthetic solution (0.25% bupivacain) under ultrasound guidance. In the intraoperative period, intravenous analgesics (dexketoprofen 50 mg, tramadol 100 mg) will be given.
  Interventions: Procedure: Serratus posterior superior intercostal plane block
- Thoracic Paravertebral Block (Active Comparator): After the patients are monitored and in the supine position, after appropriate field sterilization, a thoracic paravertebral block will be performed on the patients using 30 ml of local anesthetic solution (0.25% bupivacain) under ultrasound guidance. In the intraoperative period, intravenous analgesics (dexketoprofen 50 mg, tramadol 100 mg) will be given.
  Interventions: Procedure: Thoracic Paravertebral Block

INTERVENTIONS:
Procedure: Serratus posterior superior intercostal plane block — Serratus posterior superior intercostal plane block will be performed on the patients using 30 ml of 0.25% bupivacaine under ultrasound guidance.
  Additionally, in the postoperative period a paracetamol dose of 1 g every 8 hours and a dexketoprofen dose of 50 mg twice daily were administered iv for multimodal analgesia.
  Arms: Serratus posterior superior intercostal plane block
Procedure: Thoracic Paravertebral Block — Thoracic paravertebral block will be performed on the patients using 30 ml of 0.25% bupivacaine under ultrasound guidance.
  Additionally, in the postoperative period a paracetamol dose of 1 g every 8 hours and a dexketoprofen dose of 50 mg twice daily were administered iv for multimodal analgesia.
  Arms: Thoracic Paravertebral Block

SUMMARY:
Breast cancer is the most common malignancy in women, and surgery is one of the cornerstone treatments for breast cancer. Postoperative pain can significantly reduce patients' quality of life and acute pain may even trigger chronic pain syndrome.

Nerve blocks reduces opioid consumption in the postoperative period by providing better pain control and therefore has advantages such as fewer side effects and less risk of pulmonary and cardiac complications.

In this study; it was aimed to compare the analgesic effectiveness of serratus posterior superior intercostal plane block and thoracic paravertebral block in the postoperative period in patients who underwent mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years
* American Society of Anesthesiologists (ASA) score I-II-III
* Body Mass Index (BMI) between 18-30 kg/m2

Exclusion Criteria:

* Patients under 18 and over 80 years of age
* ASA score IV and above
* Patients with a history of bleeding diathesis
* BMI below 18 or above 30 kg/m2

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Pain Scores | On the operation day
  Pain will be assessed at rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain). Pain assessment will be done at 0st, 1st, 2nd,4th, 12th, and 24th hours after surgery.

SECONDARY OUTCOMES:
Intraoperative opioid consumption | Intraoperative period
  Remifentanil consumption for intraoperative period will be recorded
Postoperative Tramadol Consumption | On the operation day
  Tramadol consumption for 24 hours will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Yenimahalle, Ankara, Turkey (Türkiye)